CLINICAL TRIAL: NCT02575885
Title: Nicotine Delivery From Novel Non-tobacco Electronic Systems (ENDS)
Brief Title: Nicotine Delivery From Novel Non-Tobacco Electronic System in Smokers
Acronym: ENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: I 257514; NCI-2015-01187 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 257514 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH); R01DA037446 (NIH)
Record Dates: First submitted 2015-08-06; First posted 2015-10-15 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Cigarette Smoker; Current Smoker; Healthy Subject
MeSH Terms: interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (different type of ENDS product at each visit) (Experimental): Participants are asked to smoke ad lib a single cigarette of their own brand and provided with a different type of ENDS product at each visit (e-cigarette, disposable e-cigarette, eGo, personal vaporizer, e-cigar, and e-pipe) over 3.5-4 hours at least 7 days apart for 7 weeks. Participants are provided with cartridges of the same amounts of nicotine with regular (tobacco) or menthol flavor according to smoker's preference, instructed on how to use the product, asked to practice using it for 7 days, and return to the study center for their next visit.
  Interventions: Other: Electronic Cigarette; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration
- Arm II (BLU e-cigarette ENDS product with different flavors) (Experimental): Participants are asked to smoke ad lib a single cigarette of their own brand and provided with the BLU e-cigarette ENDS product with nicotine solution of one of five flavors over 3.5-4 hours at least 7 days apart for 6 weeks. Participants are provided with cartridges of maximum available amounts of nicotine and different flavors at each visit, instructed on how to use the product, asked to practice using it for 7 days, and return to the study center for their next visit.
  Interventions: Other: Electronic Cigarette; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration

INTERVENTIONS:
Other: Electronic Cigarette — Receive different type of ENDS product at each visit
  Other Names: e-Cigarette; Electronic Nicotine Delivery System
  Arms: Arm I (different type of ENDS product at each visit)
Other: Electronic Cigarette — Receive BLU e-cigarette ENDS product
  Other Names: e-Cigarette; Electronic Nicotine Delivery System
  Arms: Arm II (BLU e-cigarette ENDS product with different flavors)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies nicotine delivery from novel non-tobacco electronic system (ENDS) in smokers. Studying the levels of nicotine delivered by various types and brands of ENDS to the bloodstream, and comparing this to the levels delivered from conventional cigarettes (the participant's own brand) may help provide information about the use of nicotine-containing products that may help inform/reform current tobacco policy, practice, and harm reduction approaches.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the levels of nicotine effectively delivered by various types and brands of ENDS to the bloodstream and compare them to levels delivered from conventional cigarettes. (Study 1)

II. Explore the effect of flavorings added to nicotine solution on puffing topography and nicotine delivery and, assess and compare short-term "functional" nicotine effects of the different products by using subjective measures such as relief of craving and withdrawal symptoms. (Study 2)

SECONDARY OBJECTIVES:

I. Determine the amounts of nicotine present in various brands and types of ENDS. (Study 3)

II. Determine nicotine yields in vapors from various types of ENDS under laboratory conditions. (Study 4)

TERTIARY OBJECTIVES:

I. Develop a standardized testing protocol for ENDS that will reflect users' puffing behavior and product characteristics.

II. Develop and validate the analytical method for analysis of nicotine content in the vapor.

III. Propose a standardized puffing regimen for generating vapors for analytical purposes: Such a testing protocol will reflect the puffing behavior observed among ENDS users and should be specific to ENDS type.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I (Study 1): Participants are asked to smoke ad lib a single cigarette of their own brand and provided with a different type of ENDS product at each visit (e-cigarette, disposable e-cigarette, eGo, personal vaporizer, e-cigar, and e-pipe) over 3.5-4 hours at least 7 days apart for 7 weeks. Participants are provided with cartridges of the same amounts of nicotine with regular (tobacco) or menthol flavor according to smoker's preference, instructed on how to use the product, asked to practice using it for 7 days, and return to the study center for their next visit.

ARM II (Study 2): Participants are asked to smoke ad lib a single cigarette of their own brand and provided with the BLU e-cigarette ENDS product with nicotine solution of one of five flavors over 3.5-4 hours at least 7 days apart for 6 weeks. Participants are provided with cartridges of maximum available amounts of nicotine and different flavors at each visit, instructed on how to use the product, asked to practice using it for 7 days, and return to the study center for their next visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history
* Current moderate-to-heavy smoker as determined by:

  * Has smoked >=10 cigarettes per day regularly for the past year (by history) and (>=5 cigarettes per day Study 2 ONLY)
  * Has an expired carbon monoxide (CO) at screening visit of 8 parts per million (ppm) or more (6 ppm or more Study 2 ONLY)
* Nicotine dependence assessed as > 4 with the Fagerstrom Test for Nicotine Dependence
* Willingness to abstain from smoking for 8 hours (overnight abstinence) prior to study visits
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Unstable medical conditions (such as unstable heart disease, uncontrolled hypertension, thyroid disease, diabetes, renal or liver impairment, glaucoma, or prostatic hypertrophy) or psychiatric condition (such as current major depression, history of schizophrenia or bipolar disorder, or current regular use of psychiatric medications such as major tranquilizers and antidepressants
* Pregnancy or lactation (by history) or positive pregnancy test at screening visit
* Positive urine drug test at screening visit
* History of serious side effects from nicotine or from any nicotine replacement therapies
* Alcohol or illicit drug dependence within the past 12 months (by history and urine tests)
* Concurrent participation in another clinical trial
* Unable to communicate in English
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study intervention

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Determine Levels of nicotine effectively delivered by various types and brands of ENDS to the bloodstream and compare them to levels delivered from conventional cigarettes | Up to 1 year
  The maximum concentration of nicotine in plasma (Cmax) will be determined for each product.
Levels of nicotine effectively delivered by various types and brands of ENDS to the bloodstream and compare them to levels delivered from conventional cigarettes | Up to 1 year
  Time to maximum concentration (Tmax) will be determined for each product .
Levels of nicotine effectively delivered by various types and brands of ENDS to the bloodstream and compare them to levels delivered from conventional cigarettes | up to 1 year
  Area under the plasma concentration versus time curve (AUC) will be determined for each product.
Changes in withdrawal symptoms | up to 1 year
  Will be measured with Minnesota Withdrawal Scale
Subjective nicotine effect will be analyzed | up to 1 year
  Will be measured with Drug Effect Questionnaire
Changes in feelings and emotions | up to 1 year
  Will be measured with The Positive Negative Affect Scale

SECONDARY OUTCOMES:
Amounts of nicotine present in various brands and types of ENDS (Study 3) | Up to 1 year
  Nicotine content (mean, median, minimum and maximum) will be determined for each product
Nicotine yields in vapors from various types of ENDS under laboratory conditions (Study 4) | Up to 1 year
  Nicotine yield in vapor will be determined for each product.

OTHER OUTCOMES:
maximum concentration of nicotine in plasma (Cmax) (Study 1 and Study 2) | 2 hours post using ENDS product
  Cmax will be analyzed using a repeated measures analysis of variance, including terms for gender , race and order of treatment
The maximum concentration of nicotine in the area under the plasma concentration - time curve from 0 to 90 minutes (AUC) | 2 hours post using ENDS product
  AUC will be analyzed using a repeated measures analysis of variance, including terms for gender, race and order of treatment.
The time to maximum concentration of nicotine in plasma (tmax) | 2 hours post using ENDS product
  tmax will be analyzed using a repeated measures analysis of variance, including terms for gender , race and order of treatment
Estimated puff volume | 2 hours post using ENDS product
  Puff volume as determined with Cress Micro monitors
Estimated puff duration | 2 hours post using ENDS product
  Puff duration as determined with Cress Micro monitors

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mahoney, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Voos N, Smith D, Kaiser L, Mahoney MC, Bradizza CM, Kozlowski LT, Benowitz NL, O'Connor RJ, Goniewicz ML. Effect of e-cigarette flavors on nicotine delivery and puffing topography: results from a randomized clinical trial of daily smokers. Psychopharmacology (Berl). 2020 Feb;237(2):491-502. doi: 10.1007/s00213-019-05386-x. Epub 2019 Nov 26. PMID 31773209